CLINICAL TRIAL: NCT04519788
Title: A Double-blinded, Randomised, and Placebo-controlled Safety Study of AT-301 Nasal Spray in Healthy Adults
Brief Title: AT-301 Nasal Spray in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atossa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-301-AU-01
Record Dates: First submitted 2020-08-14; First posted 2020-08-20 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: 8 participants per cohort (randomised AT-301A/Placebo : AT-301B, 2:6). Part 1: (SAD) Participants will receive: Cohort 1 - AT- 301A/Placebo or AT-301B 0.1mL per nostril (0.2mL total); or, Cohort 2 - AT-301A/Placebo or AT-301B 0.2mL per nostril (0.4mL total).
  Part 2: (MAD) Cohort 3 - AT-301A/Placebo or AT-301B 0.1mL per nostril (0.2mL total), three times/day for 14 days; or, Cohort 4 - AT- 301A/Placebo or AT-301B) 0.2mL per nostril (0.4mL total), three times/day for 14 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AT-301B (Active Comparator): AT-301B consists of edetate disodium, glyceryl monooleate, polysorbate 80, benzalkonium chloride, microcrystalline cellulose and sodium carboxymethylcellulose (vivapur), trisodium citrate dihydrate, and purified water (HCl to adjust pH to 5.0)
  Interventions: Drug: AT-301B
- AT-301A (Placebo Comparator): AT-301A consists of sodium chloride, benzalkonium chloride and purified water (NaOH/HCl to adjust pH to 5.0)
  Interventions: Drug: AT-301A

INTERVENTIONS:
Drug: AT-301B — Nasal Spray
  Arms: AT-301B
Drug: AT-301A — Nasal Spray
  Other Names: Placebo
  Arms: AT-301A

SUMMARY:
This is a randomized, double-blind, placebo-controlled, ascending dose, multi-cohort study. The study will be conducted in 2 parts: a single ascending dose (SAD) part (Part 1) followed by a multiple ascending dose (MAD) part (Part 2).

ELIGIBILITY:
Inclusion Criteria:

Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects 2. Adult males and females, 18 to 64 years of age (inclusive) at the screening visit 3. Are non-smokers (including tobacco, e-cigarettes and marijuana) for a minimum of 1 month prior to the screening visit. Non-smokers with a significant history of smoking (> 5 pack years) are not eligible 4. Have a physically normal nasal structure (minor septum deviation allowable) 5. Body mass index (BMI) (calculated) within the range of 18 to 30 kg/m2 inclusive at the screening visit and prior to dosing on Day 1 6. Medically healthy without clinically significant abnormalities in the opinion of the investigator at the screening visit and prior to dosing on Day 1, including:

1. Physical examination without any clinically significant findings
2. Systolic blood pressure (BP) in the range of 90 to 140 mm Hg (inclusive) and diastolic BP in the range of 50 to 90 mm Hg (inclusive) after at least 5 minutes in a seated position
3. Heart rate (HR) in the range of 45 to 100 beats/min (inclusive) after at least 5 minutes rest in a semi-recumbent position
4. Normal body (tympanic) temperature (35.5 to 37.7°C, inclusive)
5. The 12-lead electrocardiogram (ECG), taken after the volunteer has been supine for at least 5 minutes, must be within normal range (corrected QT interval [QTc] males ≤450 msec; females ≤470 msec) or with abnormalities that are not hazardous to the volunteer
6. No clinically significant findings in serum chemistry, haematology, coagulation and urinalysis examinations (Note: assessed at screening only for eligibility) 7. Negative cotinine, drug and alcohol tests at screening and prior to dosing on Day 1 8. Female volunteers must:

a. Be of non-child-bearing potential i.e., have follicle-stimulating hormone levels >40 IU/L at screening and be surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before the Screening visit) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause), or b. If of childbearing potential, must have a negative pregnancy test at Screening (blood test) and before the first study drug administration (pre-dose Day 1 urine test). They must agree not to attempt to become pregnant, must not donate ova, and must agree to use a highly effective contraceptive method in addition to having their male partner use a condom (if not surgically sterilised) for penile-vaginal intercourse from signing consent until at least 30 days after the last dose of study therapy (Appendix 3) 9. Male volunteers, if not surgically sterilised, must agree not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use a condom in addition to having the female partner use a highly effective contraceptive method (Appendix 3) from signing the consent form until at least 90 days after the last dose of study therapy (Note: male volunteers are not required to use contraception with a partner of the same sex) 10. Have suitable venous access for blood sampling 11. Willing and able to comply with the requirements of the study protocol

Exclusion Criteria:

1. History or presence of the following based on self-report: of tuberculosis, asthma (including childhood asthma), severe bronchial asthma, chronic obstructive pulmonary disease, peptic ulcer or major pulmonary airway disease
2. Previous diagnoses of nasal polyps or any ear, nose and throat pathology deemed by the Investigator to affect assessment of the investigational product
3. Active hay fever, rhinitis or cold
4. History or presence of significant cardiovascular, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological or psychiatric disease, including any acute illness or surgery within the past three months determined by the PI to be clinically significant
5. Known allergy to any of the formula components
6. Current obstructive pneumonia, severe pulmonary interstitial fibrosis, alveolar proteinosis and allergic alveolitis caused by lung tumour
7. Positive serum pregnancy test for women of childbearing potential at the Screening visit or positive urine pregnancy test with confirmatory serum pregnancy test prior to dosing on Day 1
8. Females who are breastfeeding
9. Liver function test results (i.e., aspartate aminotransferase [AST], alanine aminotransferase [ALT], and gamma-glutamyl transferase [GGT]) and total bilirubin > 1.5 x fold above the upper limit of normal at the screening visit. Elevated total bilirubin allowable if an isolated finding
10. Positive testing for active human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, at the screening visit
11. Use of any prescription or over-the-counter medication (including nasal medication, herbal products, diet aids, and hormone supplements) within 7 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, except for contraceptives for female participants of childbearing potential and occasional use of paracetamol
12. Donation of blood or plasma within 30 days prior to randomization, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of study enrolment
13. Participation in another investigational clinical trial within 30 days or 5 half-lives (whichever is longer) in the case of an investigational drug prior to the first study drug administration
14. Any other condition or prior therapy, which, in the opinion of the Investigator, would make the volunteer unsuitable for this study, including unable to cooperate fully with the requirements of the study protocol or likely to be non-compliant with any study requirements

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
cardiac, pulmonary and hemodynamic parameters using 12-lead ECG | from baseline through study completion, an average of 40 days
  incidence of abnormal ECG Change from baseline in clinical laboratory parameters
  * Change from baseline in vital signs parameters
  * Change from baseline in 12-lead ECGs
  * Change from baseline in physical examination findings including auscultation
  * Change from baseline in oxygen saturation
auscultation | from baseline through study completion, an average of 40 days
  incidence of abnormal sounds Change from baseline in clinical laboratory parameters
  * Change from baseline in vital signs parameters
  * Change from baseline in 12-lead ECGs
  * Change from baseline in physical examination findings including auscultation
  * Change from baseline in oxygen saturation
determination of oxygen saturation levels | from baseline through study completion, an average of 40 days
  Incidence of abnormal oxygen saturation Change from baseline in clinical laboratory parameters
  * Change from baseline in vital signs parameters
  * Change from baseline in 12-lead ECGs
  * Change from baseline in physical examination findings including auscultation
  * Change from baseline in oxygen saturation
haematology, coagulation and serum chemistry | from baseline through study completion, an average of 40 days
  incidence of abnormal ranges Change from baseline in clinical laboratory parameters
  * Change from baseline in vital signs parameters
  * Change from baseline in 12-lead ECGs
  * Change from baseline in physical examination findings including auscultation
  * Change from baseline in oxygen saturation
urinalysis | from baseline through study completion, an average of 40 days
  incidence of abnormal measures Change from baseline in clinical laboratory parameters
  * Change from baseline in vital signs parameters
  * Change from baseline in 12-lead ECGs
  * Change from baseline in physical examination findings including auscultation
  * Change from baseline in oxygen saturation

SECONDARY OUTCOMES:
Nasal Spray Attributes Questionnaire score | from baseline through study completion, an average of 40 days
  based on a scale of 0 to 6, for each immediate attribute assessed; 0 equals none, 3 equals severe for each question; lower scores have better outcome
Incidence and severity of AE (bronchospasms) | from baseline through study completion, an average of 40 days
  AE monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Ben Canny, Study Chair — Bellberry Limited HREC
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia